CLINICAL TRIAL: NCT00097448
Title: Sudden Hearing Loss Multicenter Treatment Trial
Brief Title: Sudden Deafness Treatment Trial
Acronym: SSNHL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Steven Rauch, MD, Professor of Otology and Laryngology, Harvard Medical School, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC006296; U01DC006296 (NIH); 03-11-055 (Other: Massachusetts Eye and Ear Infirmary)
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Sudden Deafness
Keywords: sudden hearing loss; unilateral sudden sensorineural hearing loss; sudden sensorineural hearing loss; sudden unilateral hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Prednisone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Nineteen days of oral prednisone
  Interventions: Drug: prednisone
- 2 (Experimental): Four doses of methylprednisolone sodium succinate delivered by injection to the middle ear over 2 weeks
  Interventions: Drug: methylprednisolone sodium succinate

INTERVENTIONS:
Drug: prednisone — Oral, 19 days
  Arms: 1
Drug: methylprednisolone sodium succinate — Four intratympanic injections delivered to the middle ear over 2 weeks
  Arms: 2

SUMMARY:
This trial aims to compare the efficacy of oral prednisone vs. methylprednisolone injected into the middle ear for the treatment of moderate-to-severe, sudden sensorineural hearing loss (inner ear hearing loss affecting one ear that occurs over less than 72 hours).

DETAILED DESCRIPTION:
Sudden deafness is believed to affect 1:5000 people yearly. The cause is unknown. Spontaneous improvement is seen in approximately 20% of subjects. Improvement is seen in approximately 60% of subjects treated promptly with oral corticosteroids. Anecdotal case reports and uncontrolled case series have suggested the intratympanic corticosteroids may work as well or better than oral treatment. The risks of oral prednisone are well-known. In theory, intratympanic treatment should achieve a higher drug concentration at the target (inner ear) with less risk of systemic side effects. This study is a head-to-head comparison of oral prednisone vs. intratympanic methylprednisolone for primary treatment of idiopathic sudden deafness. The study is designed as a non-inferiority trial testing that hypothesis that intratympanic methylprednisolone is not inferior to oral prednisone treatment. Subjects assigned to the oral treatment arm receive 14 days of high dose prednisone (60mg/day) followed by a 5-day taper. Subjects assigned to the intratympanic treatment arm receive 4 doses of methylprednisolone injected into the middle twice weekly for two weeks. The primary outcome measure is hearing as measured by pure tone audiometry. Secondary outcomes include word recognition hearing levels and safety issues of local vs. systemic steroid side-effects and pain.

ELIGIBILITY:
Inclusion Criteria:

* Men/women 18 years and older in good health
* Unilateral sensorineural hearing loss developing within 72 hours (SSNHL)
* Pure Tone Average (PTA) (500, 1000, 2000, 4000 Hz) >/= 50 dB in the affected ear, with the affected ear >/= 30 dB worse than contralateral ear in at least one of the four frequencies
* Symmetric hearing prior to onset of SSNHL
* Hearing loss must be idiopathic
* Hearing loss must have occurred within the past 14 days
* Must be able to read or write English or Spanish

Exclusion Criteria:

SYSTEMIC DISEASE

* >21 days prior oral steroid treatment within preceding 30 days
* History of tuberculosis (TB) or positive PPD
* Insulin-dependent diabetes mellitus
* History of rheumatic disease, e.g., rheumatoid arthritis, scleroderma, lupus, etc.
* Serious psychiatric disease or psychiatric reaction to corticosteroids
* History of heart disease or transient ischemic attacks (TIAs)
* Prior treatment with chemotherapeutic or immunosuppressive drugs
* Pancreatitis
* Active peptic ulcer disease or history of gastrointestinal bleeding
* History of HIV, Hepatitis B or C
* Chronic kidney failure
* Alcohol abuse
* Active shingles
* Severe osteoporosis or non-surgical aseptic necrosis of the hip

OTOLOGIC DISEASE

* Prior history of SSNHL
* History of fluctuating hearing loss
* History of Meniere's disease
* History of chronic ear infection
* History of otosclerosis
* History of ear surgery (except childhood pressure equalization [pe] tubes)
* History of congenital hearing loss
* History of trauma immediately preceding onset of SSNHL
* History of syphilitic hearing loss
* History of genetic/hereditary hearing loss
* Skull, facial, or temporal bone anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2004-12; Primary Completion 2009-10 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rauch, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (14):
- United States (14):
  - House Ear Institute, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of Florida, College of Medicine, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Ear Institute, Farmington Hills, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - New York University School of Medicine, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Halpin C, Shi H, Reda D, Antonelli PJ, Babu S, Carey JP, Gantz BJ, Goebel JA, Hammerschlag PE, Harris JP, Isaacson B, Lee D, Linstrom CJ, Parnes LS, Slattery WH, Telian SA, Vrabec JT, Rauch S. Audiology in the sudden hearing loss clinical trial. Otol Neurotol. 2012 Aug;33(6):907-11. doi: 10.1097/MAO.0b013e31825d9a44. PMID 22805100
- [Derived] Rauch SD, Halpin CF, Antonelli PJ, Babu S, Carey JP, Gantz BJ, Goebel JA, Hammerschlag PE, Harris JP, Isaacson B, Lee D, Linstrom CJ, Parnes LS, Shi H, Slattery WH, Telian SA, Vrabec JT, Reda DJ. Oral vs intratympanic corticosteroid therapy for idiopathic sudden sensorineural hearing loss: a randomized trial. JAMA. 2011 May 25;305(20):2071-9. doi: 10.1001/jama.2011.679. PMID 21610239
- See also: Sudden Deafness — http://www.suddendeafness.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive consenting adults with SSNHL from 16 academic medical centers around the United States.
Pre-assignment Details: All subject presenting within 14 days of SSNHL onset.
Groups:
- Oral Steroids: Prednisone 60mg per day x 14 days, 5 day taper.
- Intratympanic Steroids: 1ml of methylprednisolone 10mg/ml. 4 doses over 14 days.
Period: Overall Study
Arm/Group | Oral Steroids | Intratympanic Steroids
Started | 125 | 130
Completed | 121 | 129
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Steroids | Intratympanic Steroids | Total
Number analyzed (Participants) | 125 | 130 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 130 | 255
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14) | 51 (15) | 50.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 74 | 77 | 151
Region of Enrollment [Number; unit: participants]
  United States | 122 | 127 | 249
  Canada | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Hearing Improvement
Description: Change from baseline to 2mos of 4-frequency (500, 1000, 2000, 4000Hz) pure tone average.
Time Frame: 2 months
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Oral Steroids: Prednisone
- IT Steroids: methylprednisolone
Arm/Group | Oral Steroids | IT Steroids
Number analyzed (Participants) | 121 | 129
dB | 30.7 (21.7) | 28.7 (21.5)

ADVERSE EVENTS:
Arm/Group | Oral Steroids | IT Steroids
Serious Adverse Events (participants affected / at risk) | 5/125 | 6/130
Other Adverse Events (participants affected / at risk) | 121/125 | 127/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Steroids (N=125) | IT Steroids (N=130)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Osteomyelitis of toe
Leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Bladder cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Steroids (N=125) | IT Steroids (N=130)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 70 (186)
Vertigo (Ear and labyrinth disorders) | 13 (14) | 35 (49)
Hyperglycemia (Endocrine disorders) | 36 (39) | 21 (21)
Eaer infection (Ear and labyrinth disorders) | 2 (2) | 7 (7)
Sleep disturbance (Nervous system disorders) | 44 (44) | 9 (9)
Appetite change (Endocrine disorders) | 28 (28) | 6 (7)
Tympnaic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No